CLINICAL TRIAL: NCT05534425
Title: Enhancing Innate Anti-Viral Resistance Through A Community-Based Intervention - Generation Xchange
Acronym: GenX
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Steve Cole, Ph.D., Professor of Medicine and Psychiatry & Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-001388; R01AG073053 (NIH)
Record Dates: First submitted 2022-08-31; First posted 2022-09-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Virus Infection, RNA
MeSH Terms: conditions — RNA Virus Infections

STUDY DESIGN:
Intervention Model Description: Randomized to Immediate GenX intervention vs. Waitlist Control delayed intervention
Who Masked: Investigator
Masking Description: All data collected, assayed, coded, and analyzed by researchers blind to study condition and participant identity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate GenX (Experimental): Participants immediately commence GenX program activity (intergenerational mentoring)
  Interventions: Behavioral: GenX intergenerational mentoring program
- Delayed GenX (Active Comparator): Participants engage in parallel training/educational activities, and subsequently commence GenX program activity after 3 months
  Interventions: Behavioral: GenX intergenerational mentoring program

INTERVENTIONS:
Behavioral: GenX intergenerational mentoring program — GenX trains older adults to collaborate with K-3rd grade teachers in mentoring high-need elementary school students in core reading and math skills.
  Other Names: GenX

SUMMARY:
This randomized controlled trial will test whether a recently developed community-based intergenerational mentoring program known as Generation Xchange (GenX) can enhance antiviral resistance in older African-American women and men in a low-SES urban community. Additional studies will identify the biological processes that promote resistance to respiratory virus infections and viral disease in older African-American women and men.

DETAILED DESCRIPTION:
This randomized controlled intervention trial (planned n=160) will test whether participation in the Generation Xchange (GenX) intergenerational mentoring program can reduces vulnerability to respiratory virus infections (COVID, influenzas, colds), increase antiviral immune activity (Type I interferon responses), and reduce inflammatory immune activity in older African-American women and men living in a socioeconomically disadvantaged urban community. Blood samples will also be collected to determine which biological factors are most important in protecting older African-Americans from respiratory virus infection, and which of those factors is affected by the GenX intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the GenX intergenerational mentoring program
* All GenX mentors > 50 years of age are eligible to participate in this research
* GenX program participation requires:
* Reside in neighborhood of GenX schools (South-Central Los Angeles)
* Pass basic literacy and cognitive function tests

Exclusion Criteria:

* Any health condition that would put participant at risk by enrollment/participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Concentration of Type I interferon antiviral activity (bioassay International Units / mL) | 10 months
  Blood cell production of Type I interferon activity will stimulated by exposure to a fixed dose of model viral protein (TruCulture Resiquimod R848 tubes) and quantifying Type I interferon concentration in the cell culture supernatant fluid using the standard Armstrong bioassay (Armstrong, J.A. Cytopathic effect inhibition assay for interferon: microculture plate assay. Methods in enzymology 78, 381-387 (1981).) Antiviral activity is quantified as International Units of Interferon activity / mL.

SECONDARY OUTCOMES:
Respiratory virus antibody concentration (WHO international units BAU/mL) | 10 months
  Respiratory virus infection (cold, influenza, COVID) will be assessed by multiplex IgG serological assay (MesoScale Discovery V-PLEX COVID-19 Respiratory Panel 2; https://www.mesoscale.com/products/covid-19-respiratory-panel-2-igg-k15372u/). Concentrations are quantified as WHO international Binding Antibody Units / mL.
Pro-inflammatory cytokine concentration (pg/mL) | 10 months
  Blood plasma and blood cell culture supernatant fluids will be assayed for expression of pro-inflammatory cytokines (e.g., IL1B, IL6, TNF) using the MesoScale Discovery U-PLEX Macrophage M1 Combo 1 hu assay (https://www.mesoscale.com/products/u-plex-macrophage-m1-combo-1-human-k15336k/). Measurement units are pg of cytokine / mL.

OTHER OUTCOMES:
Antiviral cell prevalence | 10 months
  Levels of key antiviral immune cells (e.g., dendritic cells, CD8+ T cells, etc.) will be assessed in blood samples by flow cytometry
Antiviral gene regulation | 10 months
  Activity of antiviral genes (RNA) and transcription factors will be assessed in blood cells
Well-being | 10 months
  Surveys will measure eudaimonic well-being and hedonic well-being
Loneliness | 10 months
  Surveys will measure loneliness, social isolation, and social support
Depressive symptoms | 10 months
  Surveys will measure symptoms of depression

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cole, Ph.D., Principal Investigator — Professor of Medicine & Psychiatry; Teresa E Seeman, Ph.D., Principal Investigator — Professor of Medicine
Locations (1):
- UCLA School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Background] Seeman T, Merkin SS, Goldwater D, Cole SW. Intergenerational mentoring, eudaimonic well-being and gene regulation in older adults: A pilot study. Psychoneuroendocrinology. 2020 Jan;111:104468. doi: 10.1016/j.psyneuen.2019.104468. Epub 2019 Sep 27. PMID 31589939